CLINICAL TRIAL: NCT07036224
Title: The Effectiveness of Training Using Exergaming on Selected Physical and Psychological Parameters in a Population of Patients Over the Age of 65 Belonging to Specific Subgroups of the Frailty Syndrome
Acronym: FREX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Frailty Exergaming KB172/2019
Record Dates: First submitted 2025-06-05; First posted 2025-06-25 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Frailty Syndrome
Keywords: frailty; older people; exergaming
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exergaming Training (Other): A 6-week standardized training program was carried out with the use of the game rehabilitation platform with Kinect sensor device. The subjects exercised under the supervision of an instructor for at least 30 minutes twice a week.
  Interventions: Device: Exergaming Training using Kinect sensor device

INTERVENTIONS:
Device: Exergaming Training using Kinect sensor device — A 6-week standardized training program was carried out with the use of the game rehabilitation platform with Kinect sensor device. The subjects exercised under the supervision of an instructor for at least 30 minutes twice a week.

SUMMARY:
This study aims to evaluate the effects of a six-week exergaming-based training program on physical and psychological parameters in individuals aged 65 and older diagnosed with frailty or pre-frailty. Participants engage in supervised exergame sessions twice weekly using the Activlife rehabilitation platform, which combines physical exercises with cognitive tasks in a virtual environment. Outcomes are assessed using validated tools including the Fried Frailty Criteria, CES-D, IPAQ-SF, Katz ADL, Lawton IADL, VES-13, Tinetti Test, and Fullerton Fitness Test. Anthropometric and functional data are collected before and after the intervention.

DETAILED DESCRIPTION:
Frailty is a clinical syndrome marked by reduced physiological reserve and increased vulnerability to adverse outcomes. Exergaming-interactive video game-based physical activity-offers a novel and potentially effective approach to counteracting physical and cognitive decline in frail older adults. While promising, existing evidence remains limited and methodologically heterogeneous.

This single-center trial investigates the effects of a six-week structured exergame training program on physical performance, functional independence, cognitive function, and mental well-being in a population of individuals aged 65+ with pre-frailty or frailty syndrome according to the Fried criteria.

Participants engage in at least 30-minute exergame-based sessions twice per week using the Activlife rehabilitation platform. The platform combines Kinect-based motion tracking with immersive therapeutic games that include physical (strength, balance, endurance) and cognitive (memory, visuospatial, logic) tasks. Sessions are supervised by a trained therapist, and game difficulty is adapted biweekly to participant capacity.

Assessments are conducted pre- and post-intervention and include: anthropometric data, frailty status (Fried criteria), depression symptoms (CES-D), physical activity (IPAQ-SF), basic and instrumental activities of daily living (Katz ADL, Lawton IADL), vulnerability (VES-13), mobility and balance (Tinetti Test), and physical fitness (Fullerton Fitness Test).

Ethical approval was obtained from the Bioethics Committee of Wroclaw Medical University (approval no. 172/2019). All participants provided written informed consent. The study adheres to the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* no medical contraindications to performing physical exercises in a standing position

Exclusion Criteria:

* diagnosed moderate or severe stage of dementia
* the presence of chronic diseases (e.g. chronic obstructive pulmonary disease, asthma, heart failure, arterial hypertension) that were uncontrolled or in an exacerbation phase

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 111 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Change in Frailty Category Based on Fried Frailty Phenotype Criteria | Baseline and through completion of exergaming training program (an average of 6 weeks)
  Frailty status will be assessed using the Fried Frailty Phenotype, which includes five criteria: unintentional weight loss, weakness (handgrip strength), slowness (gait speed), exhaustion (CES-D), and low physical activity (IPAQ-SF). Each criterion met scores 1 point (range: 0-5). Participants are classified as: robust (0 points), pre-frail (1-2 points), or frail (≥3 points). The outcome is the change in frailty category from baseline to study completion. Improvement is defined as transition to a lower-risk category (e.g., frail to pre-frail), while worsening is a shift to a higher-risk category. A decrease in frailty category indicates improvement.

SECONDARY OUTCOMES:
Frailty Score Assessed by Fried Frailty Phenotype Scale | Baseline and through completion of exergaming training program (an average of 6 weeks)
  Frailty will be assessed using the Fried frailty phenotype scale, which includes five criteria: unintentional weight loss, weakness (handgrip strength), slowness (gait speed), exhaustion (CES-D items), and low physical activity (IPAQ-SF). The score ranges from 0 to 5; higher scores indicate a worse frailty status.
Depression Symptoms Assessed by the Geriatric Depression Scale (GDS-15) | Baseline and through completion of exergaming training program (an average of 6 weeks)
  The Geriatric Depression Scale (GDS-15) includes 15 yes/no questions. Scores range from 0 to 15; higher scores indicate more severe depressive symptoms. A score ≥6 indicates increased risk of depression.
Cognitive Function Assessed by the Montreal Cognitive Assessment (MoCA) | Baseline and through completion of exergaming training program (an average of 6 weeks)
  The MoCA evaluates cognitive domains including memory, attention, and visuospatial abilities. Total score ranges from 0 to 30; higher scores indicate better cognitive function. A score below 26 suggests mild cognitive impairment.
Functional Status Assessed by the Katz Index of Independence in Activities of Daily Living (ADL) | Baseline and through completion of exergaming training program (an average of 6 weeks)
  The ADL index assesses six basic self-care activities. Scores range from 0 to 6; higher scores indicate greater independence.
Instrumental Activities of Daily Living Assessed by the Lawton-Brody Scale (IADL) | Baseline and through completion of exergaming training program (an average of 6 weeks)
  The IADL scale evaluates 8 instrumental daily tasks. Scores range from 8 to 24; higher scores indicate greater functional independence.
Physical Fitness Assessed by the Fullerton Fitness Test (Senior Fitness Test) | Baseline and through completion of exergaming training program (an average of 6 weeks)
  The Fullerton Fitness Test evaluates physical fitness in older adults across six domains.
  Chair Stand Test: number of stands in 30 seconds (lower body strength). Arm Curl Test: arm curls in 30 seconds with 2 kg (women) or 3.6 kg (men) dumbbell (upper body strength).
  Chair Sit and Reach: distance (cm) between fingertips and toes while reaching forward from a seated position (lower body flexibility).
  Back Scratch Test: distance (cm) between fingertips reaching behind the back (upper body flexibility).
  8-Foot Up and Go: time (sec) to stand, walk 2.44 m, turn, and sit (balance/agility).
  6-Minute Walk or 2-Minute Step: total distance or number of steps (aerobic endurance).
  Each test is scored separately; higher values generally indicate better fitness, except for the Up and Go test, where lower times reflect better performance.
Balance and Gait Assessed by the Tinetti Performance-Oriented Mobility Assessment (POMA) | Baseline and through completion of exergaming training program (an average of 6 weeks)
  The POMA evaluates balance and gait. Scores range from 0 to 28; scores <25 indicate risk of falling, and <19 indicate high fall risk.
Health-Related Quality of Life Assessed by the Short Form-36 (SF-36) Health Survey | Baseline and through completion of exergaming training program (an average of 6 weeks)
  The SF-36 measures quality of life across 8 domains. Scores range from 0 to 100 for each domain; higher scores indicate better perceived health.
Functional Vulnerability Assessed by the Vulnerable Elders Survey-13 (VES-13) | Baseline and through completion of exergaming training program (an average of 6 weeks)
  The VES-13 evaluates self-reported physical function and age-related risk. Scores range from 0 to 10; a score ≥3 indicates increased risk of functional decline.
Depression Symptoms Assessed by the Geriatric Depression Scale (GDS-15) | Baseline and through completion of exergaming training program (an average of 6 weeks)
  The Geriatric Depression Scale (GDS-15) is a screening tool consisting of 15 yes/no questions. Scores range from 0 to 15; higher scores indicate more severe depressive symptoms. A score of 6 or higher suggests an increased risk of depression in older adults.

CONTACTS AND LOCATIONS:
Locations (1):
- Modelowa Praktyka Lekarza Rodzinnego Maria Bujnowska-Fedak, Wroclaw, Lower Silesian Voivodeship, Poland